CLINICAL TRIAL: NCT02233491
Title: A Prospective, Randomised Controlled Trial Comparing Glycaemic Benefits of Active Versus Passive Lifestyle Intervention in Kidney Allograft Recipients
Brief Title: Comparing Glycaemic Benefits of Active Versus Passive Lifestyle Intervention in Kidney Allograft Recipients
Acronym: CAVIAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Adnan Sharif, Consultant Nephrologist, University Hospital Birmingham NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UBirminghamNHS
Record Dates: First submitted 2014-08-27; First posted 2014-09-08 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Post Transplantation Diabetes Mellitus; Obesity; Transplantation of Kidney
Keywords: PTDM; kidney transplant; lifestyle intervention; diet; exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): This group will be counselled in clinic by clinicians about the risks of glucose intolerance and will receive leaflets outlining lifestyle modification advice. The leaflets include advice on healthy eating, exercise and the importance of weight loss. However there will be no dietician referral, psychosocial intervention or focused exercise and weight loss monitoring programme. Follow up will be at routine clinic visits only where lifestyle modification advice will be reinforced as per usual clinical practise.
  Interventions: Other: Control
- Active intervention (Active Comparator): This group will receive active lifestyle modification intervention and will consist of dietician referral, graded exercise programme and weight loss advice. The dietician will be supported by Clinical Psychology services and our collaboration with a recognised expert in behavioural change therapy. The dietician will be trained with motivational interviewing skills and psychological tools will be utilised to support the active lifestyle intervention.
  Interventions: Behavioral: Active lifestyle intervention

INTERVENTIONS:
Behavioral: Active lifestyle intervention — Active intervention will comprise reviews by a renal dietician, with cognitive behaviour therapy, to provide additional support for lifestyle intervention.
  Arms: Active intervention
Other: Control — No additional support other than lifestyle advice by clinician
  Arms: Control

SUMMARY:
Post-transplantation diabetes mellitus (PTDM) is a common medical complication after kidney transplantation, related to both transplant-specific and generic risk factors, and is associated with major complications after transplantation. The current PTDM Consensus Report recommends lifestyle modification (e.g. weight loss, dietary modification, structured exercise program) as the first line therapy of choice. No recommendation is given with regards to how such guidance should be delivered. In addition no clinical evidence exists to suggest lifestyle modification provides any sustained glycaemic benefits for kidney allograft recipients.

While in the general population the benefits of lifestyle modification have been well documented with regards to attenuation of both pre-diabetic and diabetic states in the context of randomised controlled trials, no similar level of evidence exists post kidney transplantation.

This prospective randomised controlled trial is designed to compare active versus passive lifestyle intervention post kidney transplantation, to determine changes in cardio-metabolic risk profile over the course of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age>18, kidney allograft only, functioning allograft (not on dialysis), 3-24 months post-transplant

Exclusion Criteria:

* Organ transplant recipient, pre-existing diabetes, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Glucose metabolism | 6 months
  Change in insulin secretion, insulin resistance and disposition index (insulin secretion x insulin sensitivity) between baseline and post-intervention

SECONDARY OUTCOMES:
Incidence of Post-Transplantation Diabetes Mellitus | 6 months
Incidence of Impaired Glucose Tolerance | 6 months
Incidence of Impaired Fasting Glucose | 6 months
Commencement of glucose-lowering therapy | 6 months
Difference in HbA1c | 6 months
Physical changes (weight, body mass index, waist-hip ration and triceps fold thickness) | 6 months
Change in blood pressure | 6 months
Change in lipid profile | 6 months
Change in physical activity | 6 months
  Incremental Shuttle Walk Tests, Duke Activity Status Index and GP Physical Activity Questionnaire respectively
Change in psychological well-being | 6 months
  EQ5D - quality of life and health status Beck Depression Inventory (BDI-II) Situational Motivation Scale (SMS)
Change in creatinine | 6 months
Change in urine albumin-creatinine ratio | 6 months
Patient survival | 6 months and then 1-, 3-, 5- and 10-years post transplantation
  Electronic tagging to national data registries
Allograft survival | 6 months and then 1-, 3-, 5- and 10-years post transplantation
  Electronic tagging to national data registries
Hospitalization | 6 months and then 1-, 3-, 5- and 10-years post transplantation
  Electronic tagging to national data registries

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Wilcox J, Waite C, Tomlinson L, Driscoll J, Karim A, Day E, Sharif A. Comparing glycaemic benefits of Active Versus passive lifestyle Intervention in kidney Allograft Recipients (CAVIAR): study protocol for a randomised controlled trial. Trials. 2016 Aug 22;17(1):417. doi: 10.1186/s13063-016-1543-6. PMID 27550305